CLINICAL TRIAL: NCT00102596
Title: Clinical Trial Characterizing the Bioavailability of 1-Octanol in Adults With Ethanol-responsive Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050092; 05-N-0092; NCT01195909 (obsolete NCT alias)
Record Dates: First submitted 2005-01-30; First posted 2005-01-31 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Essential Tremor
Keywords: Ethanol; Alcohol Responsive; Movement Disorder; Gas Chromatography; Bioavailability; Pharmacokinetics; Essential Tremor
MeSH Terms: conditions — Essential Tremor; Movement Disorders | interventions — 1-Octanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 1-Octanol — 1-Octanol is an long-chain alcohol with potential therapeutic benefits in treating alcohol-responsive tremors based on unknown mechanisms. The intervention consisted of either 1) 1-octanol adsorbed to microcrystalline cellulose, NF (Avicel PH 102, FMC Corp., Philadelphia, PA), and fine particle silica (Sipernat 50S, Evonik Degussa Corp., Parsippany, NJ) and encapsulated in 50 mg and 250 mg dosages; or 2) a soft-gel capsule containing 1-octanol embedded in soybean oil at 50 mg and 800 mg dosages (Best Formulations Inc, City of Industry, CA).

SUMMARY:
OVERVIEW

Essential tremor (ET) is a common movement disorder affecting 0.4% of the general population and up to 14% of people 65 years and older. Response to medications such as beta blockers and primidone may be of benefit, but are often accompanied by intolerable side effects. Response to ethanol, on the other hand, has a roughly 80% chance of significant tremor reduction, though daily use of this as a treatment has potentially serious medical, social, and legal consequences.

The leading hypothesis for ET pathophysiology is an unmasking of spontaneous oscillations originating in neurons of the inferior olive. Both ethanol and 1-octanol have been shown to reduce these spontaneous oscillations in an animal model of ET; however, 1-octanol does this at a dose much lower than that leading to intoxication, suggesting in may be useful in the treatment of essential tremor. Our initial studies with 1-octanol have shown it to be safe at dosages up to 64mg/kg without signs of intoxication, while at the same time showing benefit.

OBJECTIVE

We plan to evaluate the efficacy of different 1-octanol formulations in humans based on accelerometry and spirography. We will also evaluate drug and metabolite bioavailabilities using a high performance liquid chromatography (HPLC) detection method from plasma and urine samples.

STUDY POPULATION

We will study adult subjects with ethanol-responsive Essential Tremor (ET).

DESIGN

This study is designed as a two-phase unblinded inpatient study of adults with ET receiving weight-adjusted oral dosages of 2 different formulations of 1-octanol in a crossover fashion. Phase I of the study is designed to develop an octanol detection assay using HPLC. Four subjects will receive daily escalating dosages (1-32 mg/kg) of a single 1-octanol formulation followed by a crossover trial of both formulations at a dosage of 64 mg/kg. Phase II will study 20 subjects receiving one of the two formulations at 64 mg/kg on inpatient day 1 followed by a 24 hour period of close monitoring. The second formulation will be given on day 3 and the patient will again undergo close monitoring for 24 hours.

OUTCOME MEASURES

The primary outcome measures for the study will be efficacy based on tremor ratings from accelerometry and spirography. Secondary outcome measures will be the determination of bioavailability, pharmacodynamic and pharmacokinetic profiles of octanol #61864 and octanol #68751 and their metabolites.

DETAILED DESCRIPTION:
OVERVIEW

Essential tremor (ET) is a common movement disorder affecting 0.4% of the general population and up to 14% of people 65 years and older. Response to medications such as beta blockers and primidone may be of benefit, but are often accompanied by intolerable side effects. Response to ethanol, on the other hand, has a roughly 80% chance of significant tremor reduction, though daily use of this as a treatment has potentially serious medical, social, and legal consequences.

The leading hypothesis for ET pathophysiology is an unmasking of spontaneous oscillations originating in neurons of the inferior olive. Both ethanol and 1-octanol have been shown to reduce these spontaneous oscillations in an animal model of ET; however, 1-octanol does this at a dose much lower than that leading to intoxication, suggesting it may be useful in the treatment of essential tremor. Our initial studies with 1-octanol have shown it to be safe at dosages up to 64mg/kg without signs of intoxication, while at the same time showing benefit.

OBJECTIVE

We plan to evaluate the efficacy of different 1-octanol formulations in humans based on accelerometry and spirography. We will also evaluate drug and metabolite bioavailabilities using a high performance liquid chromatography (HPLC) detection method from plasma and urine samples.

STUDY POPULATION

We will study adult subjects with ethanol-responsive Essential Tremor (ET).

DESIGN

This study is designed as a two-phase unblinded inpatient study of adults with ET receiving weight-adjusted oral dosages of 2 different formulations of 1-octanol in a crossover fashion. Phase I of the study is designed to develop an octanol detection assay using HPLC. Four subjects will receive daily escalating dosages (1-32 mg/kg) of a single 1-octanol formulation followed by a crossover trial of both formulations at a dosage of 64 mg/kg. Phase II will study 20 subjects receiving one of the two formulations at 64 mg/kg on inpatient day 1 followed by a 24 hour period of close monitoring. The second formulation will be given on day 3 and the patient will again undergo close monitoring for 24 hours.

OUTCOME MEASURES

The primary outcome measures for the study will be efficacy based on tremor ratings from accelerometry and spirography. Secondary outcome measures will be the determination of bioavailability, pharmacodynamic and pharmacokinetic profiles of octanol #61864 and octanol #68751 and their metabolites.

Addendum: Based on the results of the assays for all subjects who participated in Part 1 and 2 of this protocol, we would like to conduct an exploratory study (Part 3) consisting of two subjects receiving a dose of 128mg/kg of 1-octanol. This is meant to primarily explore the plasma concentration of 1-octanol, while also providing valuable information regarding the safety and efficacy at this higher dose. The remainder of the experimental design will be maintained, with exception of additional safety precautions which will be discussed in the protocol and consent.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with alcohol-responsive Essential Tremor
* Limb involvement should be a prominent feature of the Essential tremor
* Patients must be willing and able to safely stop and remain off any medications used to treat essential tremor for at least 4 half-lives
* Patients must be willing to abstain from ethanol and caffeine intake for at least 48 hours prior to starting the study hospitalization until study termination
* Patients must be willing and able to fast for periods of up to 12 hours during the study

EXCLUSION CRITERIA:

* Patients with abnormalities other than tremor on neurological exam
* Patients with active or past alcohol abuse or dependence
* Patients with acute or chronic severe medical conditions such as renal failure, hepatic failure or lung disease
* Patients taking primidone
* Patients on other acute or chronic medications that influence hepatic metabolism or central nervous system (CNS) function and cannot be temporarily discontinued for the length of the study
* Patients who do not wish to take a potentially intoxicating drug
* Patients with abnormalities on their baseline screening laboratory tests
* Women who are pregnant or lactating
* Patients younger than age 21
* The presence of cognitive impairment preventing informed consent or cooperation during the study
* People of Far East Asian or Native American descent, who may possess variant alleles of the genes for alcohol metabolism, i.e., alcohol dehydrogenase and aldehyde dehydrogenase, resulting in altered (slower) metabolism and potentially increased sensitivity to alcohols and their metabolites

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bikson M, Ghai RS, Baraban SC, Durand DM. Modulation of burst frequency, duration, and amplitude in the zero-Ca(2+) model of epileptiform activity. J Neurophysiol. 1999 Nov;82(5):2262-70. doi: 10.1152/jn.1999.82.5.2262. PMID 10561404
- [Background] Busenbark KL, Nash J, Nash S, Hubble JP, Koller WC. Is essential tremor benign? Neurology. 1991 Dec;41(12):1982-3. doi: 10.1212/wnl.41.12.1982. PMID 1745359
- [Background] Bushara KO, Goldstein SR, Grimes GJ Jr, Burstein AH, Hallett M. Pilot trial of 1-octanol in essential tremor. Neurology. 2004 Jan 13;62(1):122-4. doi: 10.1212/01.wnl.0000101722.95137.19. PMID 14718713
- [Background] Fahn S, Tolosa E, Marín C. Clinical rating scale for tremor. In: Jankovic J, Tolosa E, editors. Parkinson's Disease and Movement Disorders. 2nd ed. Baltimore: Williams & Wilkins; 1993. p. 225-34.
- [Result] Nahab FB, Wittevrongel L, Ippolito D, Toro C, Grimes GJ, Starling J, Potti G, Haubenberger D, Bowen D, Buchwald P, Dong C, Kalowitz D, Hallett M. An open-label, single-dose, crossover study of the pharmacokinetics and metabolism of two oral formulations of 1-octanol in patients with essential tremor. Neurotherapeutics. 2011 Oct;8(4):753-62. doi: 10.1007/s13311-011-0045-1. PMID 21594724

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Dose Escalation: Subjects fasted overnight for 6 hours and received 1, 4, 8, 16, 32 and 64 mg/kg 1-octanol at 6AM on different days. There were 2 formulations:
  1) 2 participants received 1-octanol adsorbed to microcrystalline cellulose, NF (Avicel PH 102, FMC Corp., Philadelphia, PA), and fine particle silica (Sipernat 50S, Evonik Degussa Corp., Parsippany, NJ) and encapsulated in 50 mg and 250 mg dosages; and 2) two participants received a soft-gel capsule containing 1-octanol embedded in soybean oil at 50 mg and 800 mg dosages (Best Formulations Inc, City of Industry, CA).
- Part B Then C: Fixed Dose: In Part B, subjects fasted overnight for 6 hours and received 64 mg/kg 1-octanol at 6AM of both formulations:
  1) 1-octanol adsorbed to microcrystalline cellulose, NF (Avicel PH 102, FMC Corp., Philadelphia, PA), and fine particle silica (Sipernat 50S, Evonik Degussa Corp., Parsippany, NJ) and encapsulated in 50 mg and 250 mg dosages; or 2) a soft-gel capsule containing 1-octanol embedded in soybean oil at 50 mg and 800 mg dosages (Best Formulations Inc, City of Industry, CA).
  At the completion of Parts A and B, an exploratory Part C was added in which subjects fasted overnight for 6 hours and received 128 mg/kg 1-octanol at 6AM of both formulations.
Period: Part A
Arm/Group | Part A: Dose Escalation | Part B Then C: Fixed Dose
Started | 11 | 0
Participants Assigned Treatment | 5 | 0
Completed | 4 | 0
Not Completed | 7 | 0
Not completed — Screen failures | 6 | 0
Not completed — Adverse Event | 1 | 0
Period: Part B
Arm/Group | Part A: Dose Escalation | Part B Then C: Fixed Dose
Started | 0 (Participants from Part A did not continue to Part B) | 10
Completed | 0 | 10
Not Completed | 0 | 0
Period: Part C
Arm/Group | Part A: Dose Escalation | Part B Then C: Fixed Dose
Started | 0 | 2 (Only 2 patients participated in Part C)
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline is included for all participants who passed screening and received at least 1 dose of 1-octanol, whether in Part A, B or C
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15
Height [Mean (Standard Deviation); unit: centimeters] | 169.6 (12.0)
Weight [Mean (Standard Deviation); unit: kg] | 82.9 (20.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (4.7)
Age of onset [Mean (Standard Deviation); unit: years] | 39.5 (18.6)
Disease Duration [Mean (Standard Deviation); unit: years] | 28.7 (17.2)
History of alcohol-responsive tremors [Number; unit: participants] | 15
Number of alcohol servings required for tremor response [Mean (Standard Deviation); unit: servings] — One serving of alcohol is 50 ml of 40% ethanol
  servings | 2.1 (0.3)
Family history of essential tremor [Number; unit: participants] | 13
Fahn Tolosa Marin Tremor Rating Scale [Mean (Standard Deviation); unit: scores on a scale] — Only available for the 10 participants who entered Part B. The Fahn Tolosa Marin Tremor Rating Scale was used. Minimum of this scale is 0, maximum is 164 points. Higher scores indicate more tremor. See Fahn S, Tolosa E, and Marin C (1993) "Clinical rating scale for tremor" reference provided in Protocol for full information.
  scores on a scale | 41.6 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: Normalized Mean Tremor Amplitude for Both Formulations of 64 mg/kg 1-Octanol in Part B
Description: Spirography mean tremor amplitudes were measured in the right hand of each participant at 0, 15, 30, 60, 90, 120, 150, 180, 240 and 360 minutes post-dose. Then, the scores of each participant were normalized (i.e., divided by) by their baseline tremor severity scores so that all scores are expressed as a proportion of the baseline score. Therefore, 1 is the baseline tremor severity, and lower scores indicate tremor reduction.
Time Frame: 0, 15, 30, 60, 90, 120, 150, 180, 240 and 360 minutes post-dose
Population: All participants who received both formulations of 64 mg/kg 1-octanol in Part B
Measure: Mean (Standard Error); unit: normalized score on a scale
Groups:
- 64 mg/kg 1-Octanol Cellulose-based (CEL) Formulation: Subjects fasted overnight for 6 hours. At 6AM subjects received 64 mg/kg of the 1-octanol adsorbed to microcrystalline cellulose, NF (Avicel PH 102, FMC Corp., Philadelphia, PA), and fine particle silica (Sipernat 50S, Evonik Degussa Corp., Parsippany, NJ) and encapsulated in 50 mg and 250 mg dosages.
- 64 mg/kg 1-Octanol Soybean Oil Embedded (SOY) Formulation: Subjects fasted overnight for 6 hours. At 6AM subjects received 64 mg/kg of the 1-octanol in a soft-gel capsule containing 1-octanol embedded in soybean oil at 50 mg and 800 mg dosages (Best Formulations Inc, City of Industry, CA).
Arm/Group | 64 mg/kg 1-Octanol Cellulose-based (CEL) Formulation | 64 mg/kg 1-Octanol Soybean Oil Embedded (SOY) Formulation
Number analyzed (Participants) | 10 | 10
normalized score on a scale
  Normalized score at 0 minutes | 1 (0) | 1 (0)
  Normalized score at 15 minutes post-dose | 1.009 (0.092) | 0.901 (0.181)
  Normalized score at 30 minutes post-dose | 0.826 (0.104) | 0.738 (0.132)
  Normalized score at 60 minutes post-dose | 0.786 (0.084) | 0.766 (0.171)
  Normalized score at 90 minutes post-dose | 0.670 (0.082) | 0.685 (0.16)
  Normalized score at 120 minutes post-dose | 0.662 (0.107) | 0.709 (0.119)
  Normalized score at 150 minutes post-dose | 0.680 (0.101) | 0.746 (0.143)
  Normalized score at 180 minutes post-dose | 0.645 (0.1) | 0.707 (0.113)
  Normalized score at 240 minutes post-dose | 0.791 (0.129) | 0.683 (0.112)
  Normalized score at 360 minutes post-dose | 0.894 (0.223) | 0.122 (0.098)

2. Secondary Outcome: Blood Plasma Levels of Octanoic Acid After 64 mg/kg 1-Octanol Dose
Description: Octanoic Acid is a metabolite of 1-octanol. Blood plasma levels of octanoic acid were measured at 5, 20, 45, 70, 100, 130, 160, 210, 270 and 360 minutes post-dose.
Time Frame: 5, 20, 45, 70, 100, 130, 160, 210, 270 and 360 minutes post-dose
Population: All participants who received either formulation 64 mg/kg 1-octanol in Part A or B
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 64 mg/kg 1-Octanol Cellulose-based (CEL) Formulation | 64 mg/kg 1-Octanol Soybean Oil Embedded (SOY) Formulation
Number analyzed (Participants) | 12 | 12
ng/ml
  Plasma Octanoic Acid Level at 5 min post-dose | 62.94 (29.37) | 74.16 (38.78)
  Plasma Octanoic Acid Level at 20 min post-dose | 5064.12 (4240.79) | 3885.52 (4111.65)
  Plasma Octanoic Acid Level at 45 min post-dose | 7967.97 (3078.81) | 9645.55 (5805.79)
  Plasma Octanoic Acid Level at 70 min post-dose | 6788.58 (2598.85) | 13315.26 (9162.85)
  Plasma Octanoic Acid Level at 100 min post-dose | 5701.60 (2207.62) | 9289.39 (2998.95)
  Plasma Octanoic Acid Level at 130 min post-dose | 5448.23 (1514.60) | 9605.68 (3822.29)
  Plasma Octanoic Acid Level at 160 min post-dose | 4662.88 (1719.10) | 6678.69 (2748.75)
  Plasma Octanoic Acid Level at 210 min post-dose | 3179.10 (1194.03) | 4307.74 (3135.91)
  Plasma Octanoic Acid Level at 270 min post-dose | 2248.74 (1192.60) | 2618.25 (2585.11)
  Plasma Octanoic Acid Level at 360 min post-dose | 1266.37 (822.56) | 872.51 (758.44)

3. Secondary Outcome: Heart Rate Post 1-Octanol Dose
Time Frame: 0 minutes, 15 minutes, 100 minutes and 24 hours post-dose
Population: All participants who received at least 1 dose of 1-octanol in Part A, B or C
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Groups:
- 1-Octanol Dose: Subjects fasted overnight for 6 hours. At 6AM subjects received 1-128 mg/kg of the 1-octanol
Arm/Group | 1-Octanol Dose
Number analyzed (Participants) | 15
beats per minute
  Heart Rate at 0 min | 70.8 (2.9)
  Heart Rate at 15 min | 66.6 (2.7)
  Heart Rate at 100 min | 67.1 (2.7)
  Heart Rate at 24 hours | 72.4 (2.7)

4. Secondary Outcome: PR and QTc Intervals Post 1-Octanol Dose
Time Frame: 0 minutes, 15 minutes, 100 minutes and 24 hours post-dose
Population: All participants who received at least 1 dose of 1-octanol in Part A, B or C
Measure: Least Squares Mean (Standard Error); unit: ms
Groups:
- 1-Octanol Dose: Subjects fasted overnight for 6 hours. At 6AM subjects received 1-128 mg/kg of 1-octanol
Arm/Group | 1-Octanol Dose
Number analyzed (Participants) | 15
ms
  PR Interval at 0 min | 168.8 (6.6)
  PR Interval at 15 min | 172.8 (6.2)
  PR Interval at 100 min | 171.6 (6.2)
  PR Interval at 24 hours | 168.6 (6.2)
  QTc Interval at 0 min | 433.8 (8.4)
  QTc Interval at 15 min | 436.5 (7.4)
  QTc Interval at 100 min | 433.0 (7.4)
  QTc Interval at 24 hours | 437.4 (7.5)

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | 1-octanol Dose
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-octanol Dose (N=15)
Fever (Infections and infestations) | 1 (1) — due to flu
Fall (Injury, poisoning and procedural complications) | 1 (1) — leading to fracture of one rib, accidental nature (patient slipped)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-octanol Dose (N=15)
Taste Change (Gastrointestinal disorders) | 8 (12)
Headache (General disorders) | 5 (10)
Heartburn (Gastrointestinal disorders) | 5 (7)
Gas/Bloating (Gastrointestinal disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 4 (7)
Dry Mouth (Gastrointestinal disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 3 (6)
Sedation (General disorders) | 2 (3)
Dizziness (General disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Worsening of tremor (Nervous system disorders) | 2 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Fainting (Nervous system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Dry Eyes (Eye disorders) | 1 (5)
Sweating (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment to study was ended early, as evidence became available, that a metabolite of the study substance promised significantly higher feasibility for treatment in ET.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less